CLINICAL TRIAL: NCT03525522
Title: Efficacy of Nd:Yttrium Aluminum Garnet Laser Treatment of Lichen Sclerosus
Brief Title: Nd:Yttrium Aluminum Garnet Laser Treatment for Lichen Sclerosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr Adolf Lukanovič (Other)
Collaborators: Juna d.o.o. (Industry)
Responsible Party: Sponsor-Investigator, Dr Adolf Lukanovič, Medical Director of the Division of Gynaecology, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lichen_NdYAG
Record Dates: First submitted 2018-04-05; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Lichen Sclerosus; Lichen Sclerosus Et Atrophicus
Keywords: Lichen sclerosus; laser; Nd:YAG; randomized controlled trial
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Patients assigned randomly to two groups: laser-treatment group and topical-corticosteroid group.
Who Masked: Outcomes Assessor
Masking Description: Hystology and photographic assessment performed by independant investigators unaware of the assignement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nd:YAG Laser (Experimental): Three sessions of Nd:YAG laser (1064 nm) treatment with Dynamis (Fotona, Slovenia)
  Interventions: Device: Nd:YAG Laser
- Topical Corticosteroid Diprosone (Active Comparator): Topical corticosteroid betamethasone (Diprosone, Merck Sharp & Dohme, d.o.o.) for 3 months.
  Interventions: Drug: Topical corticosteroid Diprosone

INTERVENTIONS:
Device: Nd:YAG Laser — Three sessions of Nd:YAG treatment every two weeks.
  Other Names: Nd:YAG; neodymium; Dynamis
  Arms: Nd:YAG Laser
Drug: Topical corticosteroid Diprosone — 3 months of topical corticosteroids Diprosone
  Other Names: topical corticosteroids betamethasone
  Arms: Topical Corticosteroid Diprosone

SUMMARY:
This study evaluates the efficacy of Nd:Yttrium Aluminum Garnet Laser (Nd:YAG) Treatment of Lichen sclerosus in comparison with topical corticosteroid treatment. Half of participants will receive laser treatment and the other half corticosteroid treatment and the results will be followed for 6 months.

DETAILED DESCRIPTION:
Lichen sclerosus (LS) is a chronic skin disease of unknown cause and very unpleasant symptoms which significantly influences the quality of life of the affected patients. Large majority of LS lesions is located in anogenital region where initial white flat papules usually develop into large, white patches of thin, itchy skin causing fusion of labia minora, narrowing of the introitus and burying of the clitoris. Most common symptoms are itching, pain, soreness, burning, dyspareunia and dysuria all strongly interfering with sexual function and patient's self image. Existing treatment options with systemic and topical medications (oral retinoids, topical steroids) have some drawbacks and recently the use of laser was proposed for treatment of LS. This study evaluates the safety and efficacy of Nd:Yttrium Aluminum Garnet Laser (Nd:YAG) Treatment of Lichen sclerosus in comparison with topical corticosteroid treatment. Half of participants will receive laser treatment and the other half corticosteroid treatment and the results will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed Lichen sclerosus
* voluntary signed informed consent

Exclusion Criteria:

* pregnancy
* use of photosensitizing medication
* pathology other than Lichen
* damage of tissues in the treatment area
* other inflammation
* refusal to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01-28 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual analog scale (VAS) score symptom evaluation from baseline to 3 months | Change from baseline to 3 months
  Patients will evaluate symptoms on a 0-10 VAS scale

SECONDARY OUTCOMES:
Change in Visual analog scale (VAS) score symptom evaluation from baseline to 1 month | Change from baseline to 1 month
  Patients will evaluate symptoms on a 0-10 VAS scale
Change in Visual analog scale (VAS) score symptom evaluation from baseline to 6 months | Change from baseline to 6 months
  Patients will evaluate symptoms on a 0-10 VAS scale
Comparative histological evaluation | baseline and 3 months
  biopsies taken at baseline and after treatment
patient satisfaction | 1 month
  Patients will indicate their satisfaction with the outcome of treatment on a 0-3 scale.
patient satisfaction | 3 months
  Patients will indicate their satisfaction with the outcome of treatment on a 0-3 scale.
patient satisfaction | 6 months
  Patients will indicate their satisfaction with the outcome of treatment on a 0-3 scale.
evaluation of improvement from clinical photographs | 3 months
  by blinded evaluators on a 1-4 scale

OTHER OUTCOMES:
tolerability of first laser treatment (pain and discomfort) on a 1-10 VAS scale | day 0 (first laser treatment)
  rated by patients in the laser group on a 1-10 VAS scale
tolerability of second laser treatment (pain and discomfort) on a 1-10 VAS scale | day 14 (second laser treatment)
  rated by patients in the laser group on a 1-10 VAS scale
tolerability of third laser treatment (pain and discomfort) on a 1-10 VAS scale | 1 month (third laser treatment)
  rated by patients in the laser group on a 1-10 VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Adolf Lukanović, PhD, Principal Investigator — UKC Ljubljana

IPD SHARING:
Plan to Share IPD: No